CLINICAL TRIAL: NCT03431493
Title: A Pilot, Feasibility Randomized Controlled Trial of a Behavioral Activation And Rehabilitation Intervention To Improve Psychological And Physical Impairments In Acute Respiratory Failure Survivors
Brief Title: Behavioral Activation-Rehabilitation to Improve Depressive Symptoms & Physical Function After Acute Respiratory Failure
Acronym: BEHAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00143231; K23HL138206 (NIH)
Record Dates: First submitted 2018-02-06; First posted 2018-02-13 (Actual); Results first posted 2025-09-19 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Respiratory Insufficiency; Depression; Rehabilitation; Critical Care
MeSH Terms: conditions — Respiratory Insufficiency; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral Activation - Rehabilitation (Experimental): Behavioral Activation - Rehabilitation
  Interventions: Behavioral: Behavioral Activation - Rehabilitation
- Usual Care Control (No Intervention): Usual Care Control

INTERVENTIONS:
Behavioral: Behavioral Activation - Rehabilitation — Participants will first receive a home visit from a physical therapist (PT) who will evaluate home safety and establish/verify the participant's exercise prescription. Within 1 week, an occupational therapist (OT) will visit the home to: 1) explain the purpose of behavioral activation (BA); 2) help the participant identify long-term recovery goals regarding "valued activities"; and 3) then, using the principles of BA, identify short-term goals for the next week and an action plan. The OT will then call the participant weekly (weeks 2-5) to review the status of the prior week's goals and use BA to set new goals for the upcoming week. The PT and OT will repeat home visits at week 6 to assess the participant's progress, and the OT will conduct phone calls every 2 weeks for weeks 8-12.
  Arms: Behavioral Activation - Rehabilitation

SUMMARY:
More and more people are surviving after receiving life support for respiratory failure in the intensive care unit, but these patients often experience problems with depression and physical functioning that lead to reduced quality of life. There is a lack of treatment for these patients, with past research suggesting that treatment may be more successful if mental and physical health are addressed at the same time. This research evaluates whether a therapy delivered via telephone and home visits, combining treatment for depression and physical rehabilitation, is feasible and might help patients recover.

DETAILED DESCRIPTION:
A growing number of Acute Respiratory Failure (ARF) survivors are burdened by depressive symptoms and physical impairments that last for years after intensive care unit discharge. Notably, depressive symptoms are independently associated with subsequent development of new impairments in physical functioning. There is a lack of treatment options to address these impairments in ARF survivors, with past research suggesting combining treatment for mental and physical health might be more successful.

Therefore, this study is designed to evaluate:

1. The feasibility (primary outcome) of participant recruitment and retention in a pilot randomized controlled trial (RCT) of an intervention combining Behavioral Activation (an evidence-based psychological treatment for depression) and physical rehabilitation delivered via telephone and 2 home visits over 12-weeks versus a "usual care" control group.
2. The efficacy (secondary outcome) of this Behavioral Activation-Rehabilitation intervention to reduce depressive symptoms and improve physical functioning.
3. Modifiable psychosocial risk factors for depressive symptoms in ARF survivors and the association between the intervention and these modifiable factors.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Living at home before the current admission (not in a facility)
* Acute respiratory failure managed in the ICU > 24hrs (≥1 of the following):

  1. Mechanical ventilation via an endotracheal tube or tracheostomy > 12hrs (and not ventilator-dependent before admission) OR
  2. Non-invasive ventilation (CPAP, BiPAP) > 4 hours in a 24 hour period provided for acute respiratory failure (not for Obstructive Sleep Apnoea (OSA) or other stable use) OR
  3. High flow nasal cannula with Fraction of Inspired Oxygen (FiO2) ≥ 0.5 for ≥4 hours in a 24hr period
* At least mild depressive symptoms (score ≥2 on PHQ-2 scale)

Exclusion Criteria:

* Pre-existing cognitive impairment (based on review of medical records, or proxy- administered Informant Questionnaire on Cognitive Decline in the Elderly (IQCODE) score >3.3)
* Declines informed consent or not capable of providing informed consent
* Non-English speaking
* Homelessness or living >50 miles away from study site
* Bedbound prior to the current admission
* Expected survival < 6 months according to ICU attending
* ICU Length Of Stay (LOS) > 30 days
* Not discharged home from the hospital
* Complex medical care expected soon after discharge (e.g. multiple planned surgeries, transplantation evaluation, extensive travel needs for hemodialysis, chemotherapy or radiation therapy, etc)
* Active substance abuse or psychosis
* Lack of access to telephone or inability to use telephone independently
* Pregnancy
* Suicidality
* Incarcerated

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-03-02 (Actual); Primary Completion 2024-07-18 (Actual); Study Completion 2024-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann M Parker, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Behavioral Activation - Rehabilitation | Usual Care Control
Started | 24 | 28
Completed | 21 | 26
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Behavioral Activation - Rehabilitation | Usual Care Control | Total
Number analyzed (Participants) | 24 | 28 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (14.1) | 56.0 (12.2) | 57.6 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 15 | 27
  Male | 12 | 13 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 24 | 27 | 51
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 9 | 19
  White | 14 | 18 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24 | 28 | 52

OUTCOME MEASURES:

1. Primary Outcome: Feasibility Measure Per Participant
Description: Total number of intervention visits completed per patient as a proportion of the number of intervention visits each patient is intended to complete.
Time Frame: End of intervention (12 weeks)
Population: Participants in the intervention group only
Measure: Number; unit: proportion of intended visits
Arm/Group | Behavioral Activation - Rehabilitation | Usual Care Control
Number analyzed (Participants) | 24 | 0
proportion of intended visits | 0.8 |

2. Primary Outcome: Total Feasibility Measure
Description: Total number of intervention visits completed by all study participants as a proportion of total intervention visits expected in the study
Time Frame: End of intervention (12 weeks)
Population: Participants in the intervention group only
Measure: Number; unit: proportion of total intervention visits
Units Other Than Participants: visits
Arm/Group | Behavioral Activation - Rehabilitation | Usual Care Control
Number analyzed (Participants) | 24 | 28
Number analyzed (visits) | 224 | 0
proportion of total intervention visits | 0.94 |

3. Primary Outcome: Feasibility Measure/Assess Loss to Follow-up
Description: Number of patients completing all study follow-up sessions as a proportion of the number of patients enrolled.
Time Frame: End of intervention (12 weeks)
Measure: Number; unit: proportion of participants
Arm/Group | Behavioral Activation - Rehabilitation | Usual Care Control
Number analyzed (Participants) | 24 | 28
proportion of participants | 0.88 | 0.93

4. Primary Outcome: Feasibility Measure
Description: Average number of patients enrolled per month over 12 weeks
Time Frame: End of intervention (12 weeks)
Measure: Mean (Standard Deviation); unit: average participants per month
Arm/Group | Behavioral Activation - Rehabilitation | Usual Care Control
Number analyzed (Participants) | 24 | 28
average participants per month | 0.3 (0.5) | 0.4 (0.5)

5. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS) - Anxiety Subscale
Description: An instrument used to assess anxiety symptoms. Scores range from 0 to 21. A HADS score ≥8 indicates clinically important symptoms on either subscale (more symptoms).
Time Frame: End of intervention (12 weeks)
Population: Participants with data collected
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Behavioral Activation - Rehabilitation | Usual Care Control
Number analyzed (Participants) | 21 | 26
score on a scale | 6.6 (3.6) | 6.5 (4.5)

6. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS) - Depression Subscale
Description: An instrument used to assess depressive symptoms. Scores range from 0 to 21. A HADS score ≥8 indicates clinically important symptoms on either subscale (more symptoms).
Time Frame: End of intervention (12 weeks)
Population: Participants with data collected
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Behavioral Activation - Rehabilitation | Usual Care Control
Number analyzed (Participants) | 21 | 26
score on a scale | 6.9 (4.9) | 5.0 (4.1)

7. Secondary Outcome: Personal Health Questionnaire - 8 Item Version (PHQ-8)
Description: The PHQ-8 uses a 4-point Likert scale to assess depressive symptoms. The score range is 0 to 27. Scores 5-9 indicate "mild" symptoms, 10-14 "moderate", and ≥20 "severe" depressive symptoms. Higher score more symptoms.
Time Frame: End of intervention (12 weeks)
Population: Participants with data collected
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Behavioral Activation - Rehabilitation | Usual Care Control
Number analyzed (Participants) | 19 | 25
score on a scale | 9.3 (6.9) | 6.0 (6.2)

8. Secondary Outcome: Activity Measure for Post-Acute Care Computer Adaptive Test (AMPAC-CAT) - Basic Mobility Score
Description: The AMPAC-CAT, a measure of physical function, has 269 items across three domains (basic mobility, daily activity and applied cognitive). The computer adaptive test requires a mean of 22 items from the item bank. Scores are norm-based (min 0 and mx 100). Higher scores indicate better function.
Time Frame: End of intervention (12 weeks)
Population: Participants with data collected
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Behavioral Activation - Rehabilitation | Usual Care Control
Number analyzed (Participants) | 19 | 21
score on a scale | 62.4 (8.5) | 61.4 (10.1)

9. Secondary Outcome: EQ-5D-5L - Utility Score
Description: The EQ-5D-5L is an instrument developed by the EuroQol group to measure health status. The Eq-5D-5L has 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels, ranging from 1 (no problems) to 5 (extreme problems). The resulting health utility score ranges from -0.11 to 1.00. Higher scores indicate better health status.
Time Frame: End of intervention (12 weeks)
Population: Participants with data collected
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Behavioral Activation - Rehabilitation | Usual Care Control
Number analyzed (Participants) | 21 | 26
score on a scale | 0.66 (0.31) | 0.80 (0.18)

10. Secondary Outcome: Healthcare Utilization - Readmissions
Description: Patient interview to assess the following end of study (ie ~12 weeks) variable: number of patients with inpatient readmissions
Time Frame: End of intervention (12 weeks)
Population: Patients with data collected
Measure: Count of Participants; unit: Participants
Arm/Group | Behavioral Activation - Rehabilitation | Usual Care Control
Number analyzed (Participants) | 19 | 24
Participants | 5 | 2

11. Secondary Outcome: Healthcare Utilization - Ever Utilized Mental Health Care
Description: Patient interview to assess the following end of study (ie ~12 weeks) variable: number of participants who ever utilized outpatient mental health
Time Frame: end of intervention (12 weeks)
Population: patients with data collected
Measure: Count of Participants; unit: Participants
Arm/Group | Behavioral Activation - Rehabilitation | Usual Care Control
Number analyzed (Participants) | 18 | 22
Participants | 4 | 2

12. Secondary Outcome: Healthcare Utilization - Rehabilitation
Description: Patient interview to assess the following end of study (ie ~12 weeks) variable: number of patients who ever utilized physical rehabilitation services
Time Frame: end of intervention (12 weeks)
Population: patients with data collected
Measure: Count of Participants; unit: Participants
Arm/Group | Behavioral Activation - Rehabilitation | Usual Care Control
Number analyzed (Participants) | 19 | 24
Participants | 12 | 13

13. Secondary Outcome: Behavioral Activation for Depression SCALE (BAS)
Description: This is a 25-item scale that measures changes in avoidance and activation over the course of Behavioral Activation treatment using a 7 point scale (0=not at all to 6=completely). The scale is grouped into 4 subscales (Activation, Avoidance/Rumination, Work/School Impairment, and Social Impairment). To calculate a total score, items on all subscales other than Activation are reverse-coded and then an unweighted sum is computed. Score range 0 to 150. Higher scores indicate greater activation.
Time Frame: End of intervention (12 weeks)
Population: Participants with data collected
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Behavioral Activation - Rehabilitation | Usual Care Control
Number analyzed (Participants) | 18 | 24
score on a scale | 95.3 (34.4) | 104.0 (24.8)

14. Secondary Outcome: Connor-Davidson Resilience Scale (CD RISC)
Description: This is a 25-item scale with each item rated on a 5-point scale (higher scores indicating greater resilience). The total score ranges from 0 to 100.
Time Frame: End of intervention (12 weeks)
Population: Participants with data collected
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Behavioral Activation - Rehabilitation | Usual Care Control
Number analyzed (Participants) | 18 | 25
score on a scale | 72.3 (17.0) | 78.5 (16.2)

15. Secondary Outcome: Number of Phone Attempts Needed by the OT to Reach the Participant for Each Session
Description: Measure of adherence
Time Frame: End of intervention (12 weeks)
Population: Data not collected due to COVID-19 pandemic-related changes for research staff such that fewer staff were available for research procedures, and needed to decrease burden on staff for data collection to allow for prioritizing key data elements (including primary outcomes).
Arm/Group | Behavioral Activation - Rehabilitation | Usual Care Control
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Percentage of Sessions Fully Completed and Partially Completed
Description: Measure of adherence for intervention group
Time Frame: End of intervention (12 weeks)
Population: This outcome is for intervention group only
Measure: Number; unit: percentage of sessions completed
Arm/Group | Behavioral Activation - Rehabilitation | Usual Care Control
Number analyzed (Participants) | 24 | 0
percentage of sessions completed | 0.94 |

17. Secondary Outcome: Montreal Cognitive Assessment (MoCA) - BLIND
Description: Measure of cognitive impairment. Score range 0 - 22. Higher scores indicate better cognitive function.
Time Frame: End of intervention (12 weeks)
Population: Participants with data collected
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Behavioral Activation - Rehabilitation | Usual Care Control
Number analyzed (Participants) | 20 | 24
score on a scale | 18.6 (3.4) | 17.8 (3.5)

18. Secondary Outcome: Impact of Events Scale - Revised (IES-R)
Description: This is a measure the subjective response to a specific traumatic event (in this case - critical illness and associated ICU experience). The IES-R consists of 22 items, each rated on a 5-point scale; item scores are averaged to generate a mean total score (range: 0-4). Higher score indicates more stress symptoms.
Time Frame: End of intervention (12 weeks)
Population: Participants with data collected
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Behavioral Activation - Rehabilitation | Usual Care Control
Number analyzed (Participants) | 21 | 26
score on a scale | 0.97 (0.69) | 0.85 (0.79)

19. Secondary Outcome: Brief Coping With Problems Experienced (Brief COPE) - Self Distraction Subscale
Description: A 28-item measure of coping strategies with responses provided using a 4-point Likert scale. Minimum score=2 to Maximum score=8. Higher score indicates greater use of the specified coping strategy.
Time Frame: End of intervention (12 weeks)
Population: Participants with data collected
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Behavioral Activation - Rehabilitation | Usual Care Control
Number analyzed (Participants) | 19 | 24
score on a scale | 4.8 (2.4) | 4.2 (1.7)

20. Secondary Outcome: Brief Coping With Problems Experienced (Brief COPE) - Active Coping Subscale
Description: as for outcome 19
Time Frame: End of intervention (12 weeks)
Population: Participants with data collected
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Behavioral Activation - Rehabilitation | Usual Care Control
Number analyzed (Participants) | 19 | 24
score on a scale | 5.7 (1.9) | 5.8 (2.1)

21. Secondary Outcome: Brief Coping With Problems Experienced (Brief COPE) - Denial Subscale
Description: as for outcome 19
Time Frame: end of intervention (12 weeks)
Population: Participants with data collected
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Behavioral Activation - Rehabilitation | Usual Care Control
Number analyzed (Participants) | 19 | 24
score on a scale | 3.4 (1.6) | 3.3 (2.0)

22. Secondary Outcome: Brief Coping With Problems Experienced (Brief COPE) - Substance Use Subscale
Description: as for outcome 19
Time Frame: End of intervention (12 weeks)
Population: Participants with data collected
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Behavioral Activation - Rehabilitation | Usual Care Control
Number analyzed (Participants) | 19 | 24
score on a scale | 2.1 (0.46) | 2.1 (0.45)

23. Secondary Outcome: Brief Coping With Problems Experienced (Brief COPE) - Emotional Support Subscale
Description: as for outcome 19
Time Frame: End of intervention (12 weeks)
Population: Participants with data collected
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Behavioral Activation - Rehabilitation | Usual Care Control
Number analyzed (Participants) | 19 | 24
score on a scale | 5.7 (2.2) | 6.0 (2.1)

24. Secondary Outcome: Brief Coping With Problems Experienced (Brief COPE) - Instrumental Support Subscale
Description: as for outcome 19
Time Frame: End of intervention (12 weeks)
Population: Participants with data collected
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Behavioral Activation - Rehabilitation | Usual Care Control
Number analyzed (Participants) | 19 | 24
score on a scale | 4.6 (2.2) | 5.4 (1.9)

25. Secondary Outcome: Brief Coping With Problems Experienced (Brief COPE) - Behavioral Disengagement Subscale
Description: as for outcome 19
Time Frame: End of intervention (12 weeks)
Population: Participants with data collected
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Behavioral Activation - Rehabilitation | Usual Care Control
Number analyzed (Participants) | 19 | 24
score on a scale | 3.1 (2.0) | 2.4 (1.0)

26. Secondary Outcome: Brief Coping With Problems Experienced (Brief COPE) - Venting Subscale
Description: as for outcome 19
Time Frame: End of intervention (12 weeks)
Population: Participants with data collected
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Behavioral Activation - Rehabilitation | Usual Care Control
Number analyzed (Participants) | 19 | 24
score on a scale | 4.2 (1.5) | 3.5 (1.6)

27. Secondary Outcome: Brief Coping With Problems Experienced (Brief COPE) - Positive Reframing Subscale
Description: as for outcome 19
Time Frame: End of intervention (12 weeks)
Population: Participants with data collected
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Behavioral Activation - Rehabilitation | Usual Care Control
Number analyzed (Participants) | 19 | 24
score on a scale | 5.2 (1.8) | 5.1 (2.1)

28. Secondary Outcome: Brief Coping With Problems Experienced (Brief COPE) - Planning Subscale
Description: as for outcome 19
Time Frame: End of intervention (12 weeks)
Population: Participants with data collected
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Behavioral Activation - Rehabilitation | Usual Care Control
Number analyzed (Participants) | 19 | 24
score on a scale | 5.6 (1.7) | 5.6 (2.1)

29. Secondary Outcome: Brief Coping With Problems Experienced (Brief COPE) - Humor Subscale
Description: as for outcome 19
Time Frame: End of intervention (12 weeks)
Population: Participants with data collected
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Behavioral Activation - Rehabilitation | Usual Care Control
Number analyzed (Participants) | 19 | 24
score on a scale | 3.5 (1.7) | 4.0 (2.3)

30. Secondary Outcome: Brief Coping With Problems Experienced (Brief COPE) - Acceptance Subscale
Description: as for outcome 19
Time Frame: End of intervention (12 weeks)
Population: Participants with data collected
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Behavioral Activation - Rehabilitation | Usual Care Control
Number analyzed (Participants) | 19 | 24
score on a scale | 6.6 (1.9) | 6.7 (1.5)

31. Secondary Outcome: Brief Coping With Problems Experienced (Brief COPE) - Religion Subscale
Description: as for outcome 19
Time Frame: End of intervention (12 weeks)
Population: Participants with data collected
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Behavioral Activation - Rehabilitation | Usual Care Control
Number analyzed (Participants) | 19 | 24
score on a scale | 5.3 (2.5) | 5.5 (2.4)

32. Secondary Outcome: Brief Coping With Problems Experienced (Brief COPE) - Self-Blame Subscale
Description: as for outcome 19
Time Frame: End of intervention (12 weeks)
Population: Participants with data collected
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Behavioral Activation - Rehabilitation | Usual Care Control
Number analyzed (Participants) | 19 | 24
score on a scale | 3.8 (2.0) | 3.5 (1.6)

33. Secondary Outcome: Diagnostic and Statistical Manual of Mental Disorders (DSM-5) (SCID-5)
Description: A clinical interview to assess depressive symptoms. This is a qualitative assessment.
Time Frame: End of intervention (12 weeks)
Population: Data not collected due to participant survey burden and COVID-19 pandemic-related changes for both research staff and participants.
Arm/Group | Behavioral Activation - Rehabilitation | Usual Care Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From enrollment until completion of end of intervention surveys or study drop out (4 months)
Arm/Group | Behavioral Activation - Rehabilitation | Usual Care Control
All-Cause Mortality (participants affected / at risk) | 1/24 | 2/28
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/28
Other Adverse Events (participants affected / at risk) | 0/24 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-05): https://cdn.clinicaltrials.gov/large-docs/93/NCT03431493/Prot_SAP_000.pdf